CLINICAL TRIAL: NCT03677180
Title: National Cardiogenic Shock Initiative
Acronym: NCSI
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Abiomed Inc. (Industry); Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, William W. O'Neill, Medical Director, Center for Structural Heart Disease, Henry Ford Health System
Other Study IDs: NCSI; National CSI (Other: Henry Ford Health System)
Record Dates: First submitted 2018-08-17; First posted 2018-09-19 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Heart Attack
Keywords: Cardiogenic shock; Mechanical circulatory support; National Cardiogenic Shock Initiative; Myocardial infarction; Heart attack; Acute MI; NCSI; National CSI; Impella; Shock; Hemodynamic Support
MeSH Terms: conditions — Shock, Cardiogenic; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Infarction; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the use of early mechanical circulatory support in patients presenting with acute myocardial infarction and cardiogenic shock. Patients are treated according to the National Cardiogenic Shock Initiative protocol, which emphasizes early identification of cardiogenic shock and rapid delivery of mechanical circulatory support based on invasive hemodynamics. All patients treated in this manner are enrolled in the National Cardiogenic Shock registry.

DETAILED DESCRIPTION:
Acute myocardial infarction complicated by cardiogenic shock (AMICS) is a deadly condition with a historical in-hospital survival of only 50%. To date, the only therapy proven to benefit patients in AMICS using data from randomized control trials has been early mechanical reperfusion. Accordingly, current American and European guidelines confer a class IB indication for reperfusion therapy in the setting of AMICS. Unfortunately, little progress has been made on improving survival with subsequent therapies, including intra-aortic balloon pump counter-pulsation (IABP). This lack of progress is worrisome since the incidence of AMICS appears to be increasing.

With the FDA approval of Impella (Abiomed, Danvers, MA) in AMICS, a powerful new tool has become available for hemodynamic support. Impella is a transcatheter axial flow pump, delivered percutaneous, with the ability to provide 2.5 to 4.0 liters/minute of forward flow. The device should provide sufficient forward cardiac flow to support vital organs in the majority of patients who present with AMICS. Since Impella is the only percutaneous temporary ventricular support device approved as safe and effective for use in AMICS, the use of the device has steadily grown. Unfortunately, there is little data available to providers as to the best practice patterns associated with the delivery and use of Impella in AMICS.

Using the most up-to-date research, a treatment algorithm for AMICS was developed and subsequently implemented as a quality improvement initiative throughout southeast Michigan. Patient information was gathered by each of the sites and collected in a retrospective registry. Outcomes and results were shared during quarterly meetings and concluded with a 41-patient pilot feasibility study. This initial pilot study revealed a 76% survival to discharge, a significant improvement compared to prior historical controls.

Given the promising outcomes, leaders from around the world have implemented the treatment algorithm in their local clinical practices with similar results. The investigators have therefore launched the National Cardiogenic Shock Initiative (NCSI). The aim of the NCSI is to bring together experienced centers across the nation who are experts in mechanical reperfusion therapies and have a large experience with the use of mechanical circulatory support devices to systematize care in AMICS.

Our goal is to dramatically decrease the duration patients remain in cardiogenic shock and attempt to decrease total usage and duration of vasopressors and ionotropic agents. The investigators aim to further demonstrate that rapid delivery of mechanical circulatory support will improve hemodynamics, reverse the spiraling neuro-hormonal cascade associated with cardiogenic shock, allowing clinicians to decrease use of vasopressors and inotropic agents and ultimately improve survival.

Healthcare systems that have agreed to adopt the NCSI treatment algorithm are being asked to participate in this prospective registry so that patient outcomes can be analyzed. Participating investigators will be asked to voluntarily provide data from patients completing the treatment algorithm to be included in the NCSI Registry.

ELIGIBILITY:
Registry Inclusion Criteria:

1. Symptoms of acute myocardial infarction (AMI) with ECG and/or biomarker evidence of S-T elevation myocardial infarction (STEMI) or non-S-T elevation myocardial infarction (NSTEMI)
2. Cardiogenic shock is defined as the presence of at least two of the following:

   1. Hypotension (systolic blood pressure ≤90 mm Hg, or inotropes/vasopressors to maintain systolic blood pressure ≥90 mmHg)
   2. Signs of end organ hypoperfusion (cool extremities, oliguria or anuria, or elevated lactate levels)
   3. Hemodynamic criteria represented by a cardiac index of <2.2 L/min/m2 or a cardiac power output ≤0.6 watts.
3. Patient is supported with an Impella
4. Patient undergoes PCI

Registry Exclusion Criteria:

1. Evidence of Anoxic Brain Injury
2. Unwitnessed out of hospital cardiac arrest or any cardiac arrest in which return of spontaneous circulation (ROSC) is not achieved within 30 minutes
3. IABP placed prior to Impella
4. Septic, anaphylactic, hemorrhagic, and neurologic causes of shock
5. Non-ischemic causes of shock/hypotension (pulmonary embolism, pneumothorax, myocarditis, tamponade, etc.)
6. Active bleeding for which mechanical circulatory support is contraindicated
7. Recent major surgery for which mechanical circulatory support is contraindicated
8. Mechanical complications of AMI (acute ventricular septal defect (VSD) or acute papillary muscle rupture)
9. Known left ventricular thrombus for which mechanical circulatory support is contraindicated
10. Mechanical aortic prosthetic valve
11. Contraindication to intravenous systemic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting with acute myocardial infarction and cardiogenic shock treated with mechanical circulatory support.
Sampling Method: Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W O'Neill, MD, Principal Investigator — Henry Ford Health System; Babar Basir, DO, Study Director — Henry Ford Health System
Locations (75):
- United States (75):
  - UAB Hospital, Birmingham, Alabama
  - Washington Regional Medical Center, Fayetteville, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Northwest Medical Center - Springdale, Springdale, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - St. Joseph Hospital Orange, Orange, California
  - Mercy General Hospital, Sacramento, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - St. Anthony Hospital, Lakewood, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Palmetto General Hospital, Hialeah, Florida
  - Orange Park Medical Center, Jacksonville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Elmhurst Hospital, Elmhurst, Illinois
  - Edward Hospital, Naperville, Illinois
  - Iowa Heart Center at Mercy Medical Center, Des Moines, Iowa
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - KentuckyOne Health Saint Joseph Hospital, Lexington, Kentucky
  - KentuckyOne Health Jewish Hospital, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - DMC Heart Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health Fred and Lena Meijer Heart Center, Grand Rapids, Michigan
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - Beaumont Hospital, Troy, Troy, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Research Medical Center, Kansas City, Missouri
  - SSM Health St. Louis University Hospital, St Louis, Missouri
  - CHI Health Nebraska Heart, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Englewood Hospital, Englewood, New Jersey
  - Hackensack Meridian Health Jersey Shore University Medical Center, Neptune City, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - San Juan Regional Medical Center, Farmington, New Mexico
  - Buffalo General Medical Center, Buffalo, New York
  - Mercy Hospital of Buffalo, Buffalo, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - PeaceHealth Sacred Heart Medical Center at Riverbend, Springfield, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Excela Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - North Knoxville Medical Center, Knoxville, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - Physicians Regional Medical Center, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Parkwest Regional Medical Center, Knoxville, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - Methodist Medical Center, Oak Ridge, Tennessee
  - Heart Hospital of Austin, Austin, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Methodist Hospital, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - UVA University Hospital, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Neill W, Basir M, Dixon S, Patel K, Schreiber T, Almany S. Feasibility of Early Mechanical Support During Mechanical Reperfusion of Acute Myocardial Infarct Cardiogenic Shock. JACC Cardiovasc Interv. 2017 Mar 27;10(6):624-625. doi: 10.1016/j.jcin.2017.01.014. No abstract available. PMID 28335901
- [Background] Basir MB, Schreiber TL, Grines CL, Dixon SR, Moses JW, Maini BS, Khandelwal AK, Ohman EM, O'Neill WW. Effect of Early Initiation of Mechanical Circulatory Support on Survival in Cardiogenic Shock. Am J Cardiol. 2017 Mar 15;119(6):845-851. doi: 10.1016/j.amjcard.2016.11.037. Epub 2016 Dec 18. PMID 28040188
- [Background] Basir MB, Schreiber T, Dixon S, Alaswad K, Patel K, Almany S, Khandelwal A, Hanson I, George A, Ashbrook M, Blank N, Abdelsalam M, Sareen N, Timmis SBH, O'Neill Md WW. Feasibility of early mechanical circulatory support in acute myocardial infarction complicated by cardiogenic shock: The Detroit cardiogenic shock initiative. Catheter Cardiovasc Interv. 2018 Feb 15;91(3):454-461. doi: 10.1002/ccd.27427. Epub 2017 Dec 20. PMID 29266676
- [Background] Goldberg RJ, Makam RC, Yarzebski J, McManus DD, Lessard D, Gore JM. Decade-Long Trends (2001-2011) in the Incidence and Hospital Death Rates Associated with the In-Hospital Development of Cardiogenic Shock after Acute Myocardial Infarction. Circ Cardiovasc Qual Outcomes. 2016 Mar;9(2):117-25. doi: 10.1161/CIRCOUTCOMES.115.002359. Epub 2016 Feb 16. PMID 26884615
- [Background] Kolte D, Khera S, Aronow WS, Mujib M, Palaniswamy C, Sule S, Jain D, Gotsis W, Ahmed A, Frishman WH, Fonarow GC. Trends in incidence, management, and outcomes of cardiogenic shock complicating ST-elevation myocardial infarction in the United States. J Am Heart Assoc. 2014 Jan 13;3(1):e000590. doi: 10.1161/JAHA.113.000590. PMID 24419737
- [Background] Hochman JS, Sleeper LA, White HD, Dzavik V, Wong SC, Menon V, Webb JG, Steingart R, Picard MH, Menegus MA, Boland J, Sanborn T, Buller CE, Modur S, Forman R, Desvigne-Nickens P, Jacobs AK, Slater JN, LeJemtel TH; SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. One-year survival following early revascularization for cardiogenic shock. JAMA. 2001 Jan 10;285(2):190-2. doi: 10.1001/jama.285.2.190. PMID 11176812
- [Background] Bainey KR, Armstrong PW. Transatlantic Comparison of ST-Segment Elevation Myocardial Infarction Guidelines: Insights From the United States and Europe. J Am Coll Cardiol. 2016 Jan 19;67(2):216-229. doi: 10.1016/j.jacc.2015.11.010. Epub 2015 Dec 23. PMID 26724199
- [Background] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Background] Killip T 3rd, Kimball JT. Treatment of myocardial infarction in a coronary care unit. A two year experience with 250 patients. Am J Cardiol. 1967 Oct;20(4):457-64. doi: 10.1016/0002-9149(67)90023-9. No abstract available. PMID 6059183
- [Background] Stretch R, Sauer CM, Yuh DD, Bonde P. National trends in the utilization of short-term mechanical circulatory support: incidence, outcomes, and cost analysis. J Am Coll Cardiol. 2014 Oct 7;64(14):1407-15. doi: 10.1016/j.jacc.2014.07.958. PMID 25277608
- [Result] Basir MB, Kapur NK, Patel K, Salam MA, Schreiber T, Kaki A, Hanson I, Almany S, Timmis S, Dixon S, Kolski B, Todd J, Senter S, Marso S, Lasorda D, Wilkins C, Lalonde T, Attallah A, Larkin T, Dupont A, Marshall J, Patel N, Overly T, Green M, Tehrani B, Truesdell AG, Sharma R, Akhtar Y, McRae T 3rd, O'Neill B, Finley J, Rahman A, Foster M, Askari R, Goldsweig A, Martin S, Bharadwaj A, Khuddus M, Caputo C, Korpas D, Cawich I, McAllister D, Blank N, Alraies MC, Fisher R, Khandelwal A, Alaswad K, Lemor A, Johnson T, Hacala M, O'Neill WW; National Cardiogenic Shock Initiative Investigators. Improved Outcomes Associated with the use of Shock Protocols: Updates from the National Cardiogenic Shock Initiative. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1173-1183. doi: 10.1002/ccd.28307. Epub 2019 Apr 25. PMID 31025538
- [Derived] Lorusso R. First Myocardial Resting or First Myocardial Revascularization for Cardiogenic Shock After Acute Myocardial Infarction-Related Cardiac Arrest? Still a Hamlet Dilemma...Now, With Some More Clues.... Crit Care Med. 2021 Jun 1;49(6):999-1000. doi: 10.1097/CCM.0000000000004932. No abstract available. PMID 34011835
- [Derived] Lemor A, Basir MB, Gorgis S, Todd J, Marso S, Gelormini J, Akhtar Y, Baker J, Chahin J, Abdul-Waheed M, Thukral N, O'Neill W. Impact of Age in Acute Myocardial Infarction Cardiogenic Shock: Insights From the National Cardiogenic Shock Initiative. Crit Pathw Cardiol. 2021 Sep 1;20(3):163-167. doi: 10.1097/HPC.0000000000000255. PMID 33606413
- See also: National Cardiogenic Shock Initiative Website - Henry Ford Hospital — http://www.henryford.com/cardiogenicshock

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock: Patients who presented with an acute MI (STEMI or NSTEMI) and in cardiogenic shock prior to percutaneous coronary intervention (PCI).
Period: Overall Study
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Started | 406
Completed | 406
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock: Patients who presented to the hospital with an acute MI (STEMI or NSTEMI) and in cardiogenic shock (by protocol definition) prior to percutaneous coronary intervention (PCI).
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 310
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 277
  Black | 34
  Hispanic | 28
  Other | 30
  Patient refused to reveal or information not available | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Survived at Discharge
Description: Number of Participants Who Survived at Discharge
Time Frame: through study completion (hospital discharge), an average of 30 days.
Measure: Count of Participants; unit: Participants
Groups:
- Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock: Patients who presented to the hospital with an acute MI (STEMI or NSTEMI) and in cardiogenic shock prior to percutaneous coronary intervention (PCI).
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Participants | 287

2. Secondary Outcome: Number of Participants Who Survived to 30 Days Post Hospital Discharge.
Description: Number of Participants Who Survived to 30 Days Post Hospital Discharge.
Time Frame: 30 days post-hospital discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 399
Participants | 272

3. Secondary Outcome: Number of Participants Who Survived to 1 Year Post Hospital Discharge.
Description: Number of Participants Who Survived to 1 Year Post Hospital Discharge.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 325
Participants | 173

4. Other Pre Specified Outcome: Use of MCS Pre-PCI
Description: Number of patients who receive mechanical circulatory support (MCS) pre-PCI (percutaneous coronary intervention).
Time Frame: At index Cath Lab procedure/PCI (percutaneous coronary intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Participants
  MCS placed pre-PCI | 287
  MCS placed interprocedurally | 35
  MCS placed post-PCI | 84

5. Other Pre Specified Outcome: Door to Support Time < 90 Minutes
Description: This outcome measures the time from the patient's arrival to the hospital to the time that MCS (mechanical circulatory support) was started and whether this was greater than or less than 90 minutes.
Time Frame: At index Cath Lab procedure/PCI (percutaneous coronary intervention)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Minutes | 78 [41 to 237]

6. Other Pre Specified Outcome: Number of Participants With Establishment of TIMI III Coronary Blood Flow
Description: Establishment of TIMI III (thrombolysis in myocardial infarction) coronary blood flow during index PCI (percutaneous coronary intervention) in culprit lesions.
Time Frame: At index Cath Lab procedure/PCI (percutaneous coronary intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Participants | 356

7. Other Pre Specified Outcome: Number of Vasopressors & Inotropes Used
Description: Number of vasopressor & inotropic medications being administered in patients being treated with early MCS (mechanical circulatory support) during percutaneous coronary intervention (PCI) treatment for AMICS (acute myocardial infarction with cardiogenic shock).
Time Frame: Prior to start of mechanical circulatory support during PCI (pre-PCI), post-PCI, 12-hours post-PCI, 24-hours post-PCI
Measure: Mean (Standard Deviation); unit: # of Inotropes/Vasopressors administered
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
# of Inotropes/Vasopressors administered
  # of Inotropes/Vasopressors being administered Pre-PCI | 1.0 (0.9)
  # of Inotropes/Vasopressors being administered Post-PCI | 0.9 (1.0)
  # of Inotropes/Vasopressors being administered at 12-hours Post-PCI | 1.1 (1.1)
  # of Inotropes/Vasopressors being administered at 24-hours Post-PCI | 1.0 (1.0)

8. Other Pre Specified Outcome: Average Cardiac Power Output (CPO) Measurements at Index PCI (Percutaneous Coronary Intervention), Post-PCI, 12 Hours Post-PCI, 24 Hours Post-PCI
Description: Ability to maintain a cardiac power output (CPO) measurement of > 0.6 watts.
Time Frame: At index PCI (percutaneous coronary intervention), post-PCI, 12-hours post-PCI, 24-hours post-PCI
Measure: Mean (Standard Deviation); unit: Watts (W)
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
Number analyzed (Participants) | 406
Watts (W)
  CPO pre-PCI | 0.67 (0.29)
  CPO post-PCI | 0.88 (0.44)
  CPO 12-hours post-PCI | 0.83 (0.34)
  CPO 24-hours post-PCI | 0.98 (1.32)

ADVERSE EVENTS:
Time Frame: Through study completion (hospital discharge), an average of 1 month and assessed up to 1 year post hospital discharge, up to 13 months.
Description: All 406 participants were monitored up to hospital discharge, however only 325 participants assessed for All-Cause Mortality at 1 year. Data were only available for 365 of the subjects for Adverse Events. Adverse Event Data for the remaining 41 subjects were not able to be collected by the site for adverse events. Other [non-serious] adverse events were not collected or assessed as part of the study.
Arm/Group | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock
All-Cause Mortality (participants affected / at risk) | 152/406
Serious Adverse Events (participants affected / at risk) | 83/365
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Myocardial Infarction (STEMI or NSTEMI) With Cardiogenic Shock (N=365)
Blood transfusion (Blood and lymphatic system disorders) | 83 (83) — Number of patients requiring blood transfusion during index admission.
Stroke (Vascular disorders) | 7 (7) — Number of patients with stroke reported during index admission.
Limb Ischemia (Vascular disorders) | 11 (11) — Number of patients with limb ischemia reported during index admission.

LIMITATIONS AND CAVEATS:
Given the observational nature of this study, selection bias may have contributed to the exclusion of certain patients despite aggressive measures to perform screening of consecutive patients. Similarly, reports of adverse events were self-reported without oversight or monitoring hence are prone to being under reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT03677180/Prot_000.pdf